CLINICAL TRIAL: NCT06691178
Title: Continuous Monitoring and Management of Vaginal Health Via Multifunctional OCT/OCTA/OCE Endoscopy, a Randomized Controlled Trial
Brief Title: Vaginal Changes After CO2 Laser
Acronym: OCTRCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Alma Lasers (Industry); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Felicia Lane, Division Director of Urogynecology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2080; 1R01EB030558-01A1 (NIH)
Record Dates: First submitted 2024-09-04; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Genitourinary Syndrome of Menopause
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CO2 Vaginal Laser treatment (Experimental): Laser treatment with a Fractional/Pixel CO2 laser (Femilift, Alma Lasers) will be performed with the following settings and procedure: single pulse; first pass 50-100 millijoules/pixel of energy, and 50-100 millijoules/pixel for the second pass. The energy level will be adjusted within the range based on the subject's comfort level. The same procedures will be followed for the sham group but no pulse will be generated.
  Interventions: Diagnostic Test: Optical coherence tomography (OCT)
- Sham - no vaginal laser treatment (Sham Comparator): The vaginal laser probe will be placed as usual but no energy will be delivered to the tissue.
  Interventions: Diagnostic Test: Optical coherence tomography (OCT)

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography (OCT) — The OCT device with cover will be used to take measurements at four areas in the vaginal canal: the proximal posterior aspect, proximal anterior, distal anterior, and distal posterior. The proximal and distal points will be marked on the OCT cover during the first set of measurements. Markings will be used to guide measurements during subsequent visits.

SUMMARY:
Genitourinary syndrome of menopause (GSM) occurs due to a decline in estrogen levels as a woman approaches menopause. The syndrome negatively impacts women's quality of life and is characterized by vaginal dryness, burning, diminished lubrication, painful intercourse and urinary symptoms such as frequency and urgency. GSM is diagnosed by symptom assessment and physical exam, with current mainstay of treatment being vaginal estrogen. Women with a history of breast cancer, gynecologic cancer, or venous thromboembolism may not be candidates for hormonal therapy. Thus, there has been a quest for effective non-hormonal forms of treatment for GSM. The use of vaginal CO2 laser treatment for GSM has shown promising results.

In this study, we aim to use long-wavelength optical coherence tomography/angiography/elastography (OCT/OCTA/OCE) to document changes that occur in the vaginal epithelium during menopause as well as after treatment for GSM. OCT is a well-studied technology and is widely used in Dermatology and Ophthalmology. In collaboration with the Beckman Laser Institute (BLI), we have developed a non-invasive vaginal probe (HS# 2017-3686). The probe has subsequently been used in previous studies to validate measurements in the vaginal epithelium (HS# 2019-5446). A previous RCT compared clinical response to laser therapy to a control group that received a low level of laser therapy. The study also did not examine histology. This will be a randomized controlled trial in which women will be enrolled into one group receiving laser therapy and compared to a true sham group that will not receive laser therapy at all. Response will be measured primarily by OCT device as well as optional vaginal biopsies. There will also be questionnaires and exam of the vaginal tissue using the VHI.

DETAILED DESCRIPTION:
Genitourinary Syndrome of Menopause (GSM) is a broad term that describes symptoms that arise from a physiologic decline in estrogen levels. Although GSM is not a life-threatening condition, it has a negative impact on a woman's quality of life with regards to general health and sexual function. Considering the years after menopause can make up the longest portion of a woman's life, safe and effective therapies to relieve the progressive menopausal symptoms over a long period are needed. Hormone therapy is commonly used to supplement the body's natural estrogen and relieve menopause symptoms. However, safety concerns associated with long-term hormone therapy exists, including the increased risk of blood clots, breast cancer, and endometrial cancer. An alternative treatment approach has been recently proposed for the relief of menopausal symptoms based on an energy-based device. While laser therapy, like CO2 micro-ablation, has demonstrated clear benefits in dermatology, it is a new application in female pelvic medicine with limited long-term follow-up.

For benign conditions such as GSM, an invasive biopsy is not indicated and not standard of care. But without histologic information, the complete pathophysiology of GSM and how alternative treatment options such as fractional-CO2 laser therapy may work, remain poorly understood. Thus, a non-invasive tool that can obtain tissue histopathological information before and over the time course of treatment is lacking in the field of pelvic medicine. We have already developed and optimized a vaginal OCT/OCTA/OCE imaging system (HS# 2017-3686) that can be used in women [9]. This technology is able to obtain a comprehensive image of the vaginal epithelium, blood vessels, and lamina propria using 1.7 μm or 1.3 μm OCT, OCTA, and OCE. In the HS# 2019-5446 IRB study, we measured the the VET (vaginal epithelium thickness) and BVD (blood vessel density) changes in four vaginal locations: distal anterior and posterior and proximal anterior and posterior at each visit using the OCT device. We saw improvement in the in the mean difference in the VET and BVD at each visit compared to the baseline measurements at visit 1. These measurements reached statistical significance by visit 4.

The focus of this study is to compare vaginal laser therapy to a sham group using the objective measurements the OCT device can provide. We expect the vaginal epithelium thickness and blood vessel density to be statistically significantly improved by the fourth follow-up visit after three laser treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Birth sex: female
2. Desire for vaginal laser therapy for GSM
3. Age >=18 years old
4. Willingness to forego other treatments for GSM within the study period
5. Diagnosed as postmenopausal (either by surgical removal of ovaries or natural progression defined as no periods in 1 year)

Exclusion Criteria:

1. History of pelvic radiation
2. On hormone replacement therapy in the prior 3 months
3. Not able or willing to follow study instructions
4. Current diagnosis of recurrent UTIs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal epithelial thickness | Measurements will be obtained once a month for the first three months. Measurements will be obtained at subsequent follow up visits every 3 months for 1 year.
  OCT measurement of vaginal epithelial thickness
Blood vessel density | Measurements will be obtained once a month for the first three months. Measurements will be obtained at follow up visits every 3 months for 1 year.
  OCT measurement of blood vessel density

SECONDARY OUTCOMES:
Vulvovaginal symptoms questionnaire (VSQ) | Questionnaire will be obtained at baseline, during each treatment visit (once a month) and each follow up visit (every 3 months for 1 year).
  Validated questionnaire to assess genitourinary syndrome of menopause symptom severity in postmenopausal patients. The score is from 0-20. Higher scores indicate worse symptoms.
Vaginal health index (VHI) | Physical exam will be performed at baseline, during each treatment visit (once a month) and each follow up visit (every 3 months for 1 year).
  Scoring system based on provider physical exam assessing optimization of vaginal health. Scores are from 5-25, higher scores indicate better vaginal health.
Vaginal Microbiome | A vaginal swab will be obtained at baseline, during each treatment visit (once a month) and each follow up visit (every 3 months for 1 year).
  Vaginal swab
Patient Global Impression | Questionnaire will be completed starting the second treatment visit (once a month) and each follow up visit (every 3 months for 1 year).
  Single item questionnaire assessing subjective improvement on a likert scale.
Assessment of Quality of Life 6D | Measurements will be obtained once a month for the first three months. Measurements will be obtained at subsequent follow up visits every 3 months for 1 year.
  Validated questionnaire assessing quality of life. The scores range from 20 - 99 points.

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Lane, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Beckman Laser Institute, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with anyone outside of the study group

REFERENCES:
- [Background] Gandhi J, Chen A, Dagur G, Suh Y, Smith N, Cali B, Khan SA. Genitourinary syndrome of menopause: an overview of clinical manifestations, pathophysiology, etiology, evaluation, and management. Am J Obstet Gynecol. 2016 Dec;215(6):704-711. doi: 10.1016/j.ajog.2016.07.045. Epub 2016 Jul 26. PMID 27472999
- [Background] Diedrich CM, Kastelein AW, Verri FM, Weber MA, Ince C, Roovers JWR. Effects of topical estrogen therapy on the vaginal microcirculation in women with vulvovaginal atrophy. Neurourol Urodyn. 2019 Jun;38(5):1298-1304. doi: 10.1002/nau.23977. Epub 2019 Apr 4. PMID 30947367
- [Background] Santoro N, Komi J. Prevalence and impact of vaginal symptoms among postmenopausal women. J Sex Med. 2009 Aug;6(8):2133-42. doi: 10.1111/j.1743-6109.2009.01335.x. Epub 2009 Jun 1. PMID 19493278
- [Background] Qiu S, Arthur A, Jiang Y, Miao Y, Li Y, Wang J, Tadir Y, Lane F, Chen Z. OCT angiography in the monitoring of vaginal health. APL Bioeng. 2023 Nov 7;7(4):046112. doi: 10.1063/5.0153461. eCollection 2023 Dec. PMID 37946874
- [Background] Pitsouni E, Grigoriadis T, Falagas ME, Salvatore S, Athanasiou S. Laser therapy for the genitourinary syndrome of menopause. A systematic review and meta-analysis. Maturitas. 2017 Sep;103:78-88. doi: 10.1016/j.maturitas.2017.06.029. Epub 2017 Jun 27. PMID 28778337
- [Background] Athanasiou S, Pitsouni E, Antonopoulou S, Zacharakis D, Salvatore S, Falagas ME, Grigoriadis T. The effect of microablative fractional CO2 laser on vaginal flora of postmenopausal women. Climacteric. 2016 Oct;19(5):512-8. doi: 10.1080/13697137.2016.1212006. Epub 2016 Aug 24. PMID 27558459
- [Background] Tadir Y, Gaspar A, Lev-Sagie A, Alexiades M, Alinsod R, Bader A, Calligaro A, Elias JA, Gambaciani M, Gaviria JE, Iglesia CB, Selih-Martinec K, Mwesigwa PL, Ogrinc UB, Salvatore S, Scollo P, Zerbinati N, Nelson JS. Light and energy based therapeutics for genitourinary syndrome of menopause: Consensus and controversies. Lasers Surg Med. 2017 Feb;49(2):137-159. doi: 10.1002/lsm.22637. Epub 2017 Feb 21. PMID 28220946
- [Background] Li FG, Maheux-Lacroix S, Deans R, Nesbitt-Hawes E, Budden A, Nguyen K, Lim CY, Song S, McCormack L, Lyons SD, Segelov E, Abbott JA. Effect of Fractional Carbon Dioxide Laser vs Sham Treatment on Symptom Severity in Women With Postmenopausal Vaginal Symptoms: A Randomized Clinical Trial. JAMA. 2021 Oct 12;326(14):1381-1389. doi: 10.1001/jama.2021.14892. PMID 34636862
- [Background] Li Y, Sudol NT, Miao Y, Jing JC, Zhu J, Lane F, Chen Z. 1.7 micron optical coherence tomography for vaginal tissue characterization in vivo. Lasers Surg Med. 2019 Feb;51(2):120-126. doi: 10.1002/lsm.23003. Epub 2018 Jul 30. PMID 30058722
- [Background] Chang CH, Myers EM, Kennelly MJ, Fried NM. Optical clearing of vaginal tissues, ex vivo, for minimally invasive laser treatment of female stress urinary incontinence. J Biomed Opt. 2017 Jan 1;22(1):18002. doi: 10.1117/1.JBO.22.1.018002. PMID 28301637